CLINICAL TRIAL: NCT02228837
Title: The Health-Promoting Role of Pears in Men and Women With Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Pear Bureau Northwest (Unknown); Washington Tree Fruit Research Commission (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bahram Arjmandi, Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RF02456
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 12 weeks of consuming 50 g pear-flavored placebo powder mixed with 480 ml per day (1/2 in the morning and 1/2 in the evening at least 6-8 hours apart).
  Interventions: Dietary Supplement: Placebo
- Pear (Experimental): 12 weeks of consuming 2 medium-sized pears per day (1 in the morning and 1 in the evening at least 6-8 hours apart).
  Interventions: Dietary Supplement: Pear

INTERVENTIONS:
Dietary Supplement: Pear
  Arms: Pear
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The hypothesis of this study is that the daily consumption of 2 medium-sized pears for twelve weeks will improve blood pressure, lipid profiles, glycemic control and insulin resistance, inflammatory and oxidative status in men and women with metabolic syndrome. 50 men and women between the ages of 45 and 65 who have three of the five features of metabolic syndrome as defined by the Adult Treatment Panel III will be included in the study. After a two-week run-in phase, eligible men and women will be randomly assigned to one of two treatment groups: 1) 2 medium-sized pears; or 2) 50 g placebo powder daily for twelve weeks. After an initial telephone screening, all participants will be requested to report to the study site for their first visit. On the first visit (screening), participants will be provided with verbal and written explanation of the project. They will then be asked to sign an informed consent form, followed by measuring waist circumference, resting brachial blood pressure, fasting serum triglycerides, high density lipoprotein cholesterol, and glucose levels to confirm metabolic syndrome. Baseline assessments will be performed for medical history, medication use, dietary intake, and physical activity. Qualified participants will be scheduled for their second visit two weeks later (actual baseline data collection) and randomly assigned to their treatment group. On the second (baseline) visit between the hours of 6-11 A.M., blood pressure will be measured followed by blood draw and urine collection. Anthropometrics and body composition will be measured. Questionnaires regarding diet, physical activity, and gastrointestinal health will be performed. Participants will be provided with their assigned treatment and will receive standard instructions on how to fill out daily diaries for their treatment. All assessments will be repeated at 6- (third visit), and 12-week (final visit) intervals. All assessments and information will be collected after an overnight fast and 12 hours after the abstinence of caffeine and/or 24 hours after the last bout of moderate to heavy physical activity. After the initial 12 weeks, participants will undergo a 4-week washout period in which they will not consume either the intervention or the placebo. After the 4-week washout period, participants will crossover into the other group to receive either the intervention or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 45-65 years old
* Three of the following five features at the screening visit:
* Waist circumference of ≥ 40 inches for men and 35 inches for women
* Serum triglycerides ≥ 150 mg/dL
* Serum high density lipoprotein cholesterol levels < 40 mg/dL for men and <50 mg/dL for women
* Blood pressure ≥ 130/85 mm Hg
* Fasting blood glucose level ≥ 110 mg/dL

Exclusion Criteria:

* Taking hypoglycemic, antihypertensive or cholesterol-lowering medications
* Diagnosed cardiovascular disease
* Uncontrolled hypertension (≥ 160/100 mmHg)
* Diabetes mellitus
* Other active chronic diseases such as cancer, asthma, glaucoma, thyroid, kidney, liver and pancreatic disease
* Participating in a weight loss program
* Heavy smokers (> 20 cigarettes per day)
* Heavy drinkers (> 12 alcoholic drinks per week)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  By measuring brachial blood pressure at rest.

SECONDARY OUTCOMES:
Atherogenic Markers | 12 weeks
  By measuring lipid profiles and atherogenic risk ratios.
Inflammation | 12 weeks
  By measuring markers of inflammation.
Oxidative Stress | 12 weeks
  By measuring markers of oxidative stress.
Insulin Sensitivity | 12 weeks
  By measuring fasting glucose, insulin, homeostatic model of insulin resistance, and hemoglobin A1C.
Body Composition | 12 weeks
  By measuring fat mass and fat-free mass using dual-energy X-ray absorptiometry and anthropometrics.
Gastrointestinal Health | 12 weeks
  By using a validated Seven-Day Bowel Movement Questionnaire and serum levels of short-chain fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Bahram H. Arjmandi, PhD, RD, Principal Investigator — Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University; Sarah A. Johnson, PhD, RDN, Principal Investigator — Department of Food Science and Human Nutrition, Colorado State University
Locations (1):
- Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Navaei N , Pourafshar S , Akhavan NS , Litwin NS , Foley EM , George KS , Hartley SC , Elam ML , Rao S , Arjmandi BH , Johnson SA . Influence of daily fresh pear consumption on biomarkers of cardiometabolic health in middle-aged/older adults with metabolic syndrome: a randomized controlled trial. Food Funct. 2019 Feb 20;10(2):1062-1072. doi: 10.1039/c8fo01890a. PMID 30720034